CLINICAL TRIAL: NCT05056350
Title: Professional Life After Breast Cancer: Feasibility of a Coaching Program for an Adapted Return to Work
Acronym: VISIBILITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2020-07 VIS; 2020-A00955-34 (Other: ID RCB number of competent autority in France)
Record Dates: First submitted 2021-09-07; First posted 2021-09-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: return to work
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of the feasibility and impact of a back-to-work support program (Other): questionnaires, back to work coaching
  Interventions: Other: Questionnaires; Other: back to work coaching

INTERVENTIONS:
Other: Questionnaires — Quality of life questionnaires, work perception questionnaires, psychological distress questionnaire
Other: back to work coaching — Back-to-work support program including an individual interview to identify patient needs and expectations, 7 coaching workshops (every 3 weeks +/- 15 days) and a final individual assessment post workshops

SUMMARY:
The diagnosis of breast cancer and the treatments implemented have a significant impact on the professional situation.

Maintaining employment and/or reintegration into working life are therefore major issues for cancer patients.

This trial proposes to study the feasibility of a support/coaching program for a return to work in patients after breast cancer.

DETAILED DESCRIPTION:
This study involves patients with breast cancer at the end of their adjuvant treatment.

The aim of this study is to evaluate the feasibility of a support program for an adapted return to work of these patients.

This back-to-work support program including an individual interview to identify patient needs and expectations, 7 coaching workshops (every 3 weeks +/- 15 days) and a final individual assessment post workshops.

The evolution of quality of life, psychological distress and perceptions concerning work will also be evaluated through assessments and questionnaires before (inclusion) and after the support program [1 month (+/- 7 days) and 6 months (+/- 1 month) after the final individual assessment].

The study also aims to estimate the recruitment rate in the study and to assess the satisfaction of this support program.

Finally, the impact of this support program on the return to work will be described.

This initial study will eventually lead to a larger research protocol on the effectiveness of the program, using a randomized controlled trial design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients cared at the Montpellier Cancer Institute (ICM) for non-metastatic breast cancer who have received adjuvant treatment (radiotherapy and/or chemotherapy)
* Patient who has completed adjuvant treatment, except for hormonotherapy
* Patient practicing a profession at the time of diagnosis, looking for a job or in professional retraining at the time of diagnosis
* Patient expressing spontaneously or on request of the oncologist physical or psychological difficulties in the professional field
* Patient wishing to be accompanied for an adapted return to her current job or for a return to a new more adapted job
* Patient who signed the informed consent after informed information by her clinician

Exclusion Criteria:

* Metastatic breast cancer or any other cancer within the last 5 years
* Patient who haven't completed herr adjuvant treatment (chemotherapy and/or radiotherapy)
* Psychological condition requiring therapeutic support (objectified by the Mini International Neuropsychiatric Interview test (MINI) by identifying a Diagnostic and Statistical Manual (DSM)-IV Axis I psychiatric disorder (American Psychiatric Association, 1994) Sheehan et al., 1998) with the patient's refusal of adequate psychiatric treatment (medicated or not) at the time of inclusion in the study
* Severely impaired global cognitive functioning (objectified by an adjusted score of less than 20 on the Montreal Cognitive Assessment (MoCA) test)
* Physical inability to answer questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Patient adherence of a coaching program for an adapted return to work | through study completion, an average of 1 year
  Assessment of the feasibility of a support program for an adapted return to work in patients with breast cancer, after their adjuvant treatment. Feasibility is defined by the proportion of patients who have adhered to the support program, with the patient attending at least 5 of the 7 proposed sessions.

SECONDARY OUTCOMES:
Impact of the support program on the return to work | At 1 month and at 6 months
  Description of the impact of the support program on return to work, defined as any return to work, regardless of the number of hours worked by the patient before diagnosis. The description will be made by the number of patients with a return to work (resumption of previous activity or new professional activity) and, if applicable, at what date.
Estimation of recruitment rate in the study | At inclusion
  Estimation of recruitment rate in the study by the proportion of patients agreeing to participate in the program among eligible patients
Evolution of perceptions regarding work importance | AT inclusion, at 1 month and 6 months
  The score on a visual analog "work importance" scale, ranging from 0 to 10 (10 indicating a high level of importance).
Evolution of Work Ability | AT inclusion, at 1 month and 6 months
  by the Work Ability Index, on a scale of 0 to 10 (10 indicating significant ability).
Evolution of self-efficacy | AT inclusion, at 1 month and 6 months
  The self-efficacy score , obtained on the Lagerveld et al. (2010) to 11 items (with a high score indicating a high degree of self-efficacy.
Satisfaction of the support program Satisfaction of the support program | At 1 month and at 6 months
  Assessment of the satisfaction of the support program by coaching. Assessment by program satisfaction score on a visual analog scale ranging from 1 to 10 (10 indicating high satisfaction)
Quality of life (QoL) | At inclusion, at 1 month and at 6 months
  By the QoL score obtained on the EORTC QLQ-C30 & EORTC QLQ-BR23 questionnaires
Evolution of the psychological distress of patients | At inclusion, at 1 month and at 6 months
  Description of the evolution of the psychological distress of patients. Measured by HADS scale (Hospital Anxiety and Depression Scale). The HADS is a 14 items questionnaire: 7 items related to anxiety and 7 items related to depression scored on a scale. Scores for items in each subscale of the HADS are summed to produce an anxiety score (HADS-A) or a depression score (HADS-D), or can be added to produce a total score corresponding to emotional distress (HADS-T). Each item is rated on a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), for a total score ranging from 0-21 for each subscale. The entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Guerdoux, Dr, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Institut du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arfi A, Baffert S, Soilly AL, Huchon C, Reyal F, Asselain B, Neffati S, Rouzier R, Hequet D. Determinants of return at work of breast cancer patients: results from the OPTISOINS01 French prospective study. BMJ Open. 2018 May 18;8(5):e020276. doi: 10.1136/bmjopen-2017-020276. PMID 29776920
- [Background] Banning M. Employment and breast cancer: a meta-ethnography. Eur J Cancer Care (Engl). 2011 Nov;20(6):708-19. doi: 10.1111/j.1365-2354.2011.01291.x. Epub 2011 Sep 20. PMID 21933291
- [Background] Barnes AJ, Robert N, Bradley CJ. Job attributes, job satisfaction and the return to health after breast cancer diagnosis and treatment. Psychooncology. 2014 Feb;23(2):158-64. doi: 10.1002/pon.3385. Epub 2013 Sep 3. PMID 24000141
- [Background] de Boer AG, Verbeek JH, Spelten ER, Uitterhoeve AL, Ansink AC, de Reijke TM, Kammeijer M, Sprangers MA, van Dijk FJ. Work ability and return-to-work in cancer patients. Br J Cancer. 2008 Apr 22;98(8):1342-7. doi: 10.1038/sj.bjc.6604302. Epub 2008 Mar 18. PMID 18349834
- [Background] Ekbladh E, Thorell LH, Haglund L. Perceptions of the work environment among people with experience of long term sick leave. Work. 2010;35(2):125-36. doi: 10.3233/WOR-2010-0964. PMID 20164607